CLINICAL TRIAL: NCT00566345
Title: Double Blind, Placebo Controlled Phase 3 Study of the Efficacy of an Investigational Vero Cell-Derived Influenza Vaccine (VCIV) to Prevent Culture Confirmed Influenza Infection (CCII)
Brief Title: Efficacy Study of an Investigational Influenza Vaccine (Vero Cell Derived) to Prevent Culture Confirmed Influenza Infection (CCII)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 720703
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Results first posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-07

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Influenza vaccine (Experimental): Vero-cell derived influenza vaccine
  Interventions: Biological: Inactivated seasonal influenza vaccine (split virus, Vero cell-derived)
- Placebo (Placebo Comparator): Phosphate buffered saline (packaged in syringes identical to those used for the investigational vaccine)
  Interventions: Other: Phosphate buffered saline

INTERVENTIONS:
Biological: Inactivated seasonal influenza vaccine (split virus, Vero cell-derived) — Trivalent, non-adjuvanted vaccine; dose: 0.5 ml
  Arms: Influenza vaccine
Other: Phosphate buffered saline — Packaged in syringes identical to those used for the investigational vaccine; dose: 0.5 ml
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to demonstrate the efficacy of an investigational Vero-cell derived influenza vaccine to prevent infection in an adult population with an influenza virus that is antigenically similar to one of the three strains in the vaccine. All subjects will be randomized to receive a single 0.5 ml intramuscular injection from one of three lots of seasonal Vero-cell derived influenza vaccine or saline placebo. Subjects will be monitored for 180 days following vaccination for occurrence of adverse events. For determining antibody response, subjects will have one blood draw before and one blood draw 21 days after vaccination.

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects who

* are 18 to 49 years of age, inclusive, on the day of screening
* have an understanding of the study, agree to its provisions and give written informed consent prior to study entry
* If female and capable of bearing children - have a negative urine pregnancy test result within 24 hours of the vaccination on Study Day 0 and agree to employ adequate birth control measures. For the purposes of this study adequate birth control measures incorporate two types of the following FDA approved birth control measures through 60 days after the vaccination: hormonal types of birth control (such as implants, birth control pills, patches or other methods) or an intrauterine device, OR an additional barrier type of birth control measure (i.e., condoms, diaphragms, cervical caps, etc.).

Exclusion Criteria:

Subjects who have any of the risk factors for complications from influenza infection as defined by the Centers for Disease Control and Prevention (CDC):

* pregnancy
* chronic disorders of the pulmonary or cardiovascular system including asthma (hypertension is not considered a high risk condition)
* chronic renal disorders
* chronic hepatic disorders
* chronic hematological disorders
* chronic metabolic disorder (including diabetes mellitus)
* immunosuppression (including immunosuppression caused by medications or HIV)
* any condition that can compromise respiratory function or the handling of respiratory secretions or that can increase risk for aspiration (e.g., cognitive dysfunction, spinal cord injuries, seizure disorders or other neuromuscular disorders)
* residence in a nursing home or other chronic care facility that houses persons of any age who have chronic medical conditions
* household contact with children aged 0 to 59 months or of someone who is included in the risk categories listed above
* employment as a health care worker

Subjects are also excluded if they

* are unable to lead an independent life as a result of either physical or mental handicap
* have a history of severe allergic reactions or anaphylaxis
* have an oral temperature of >= 99.5° F (37.5°C) on the day of vaccination in this study. [NOTE: Subjects meeting this exclusion criterion may be rescheduled for vaccination and study entry at a later date provided: 1.) oral temperature has decreased to < 99.5°F (37.5°C) on rescheduled date, 2.) all other inclusion/exclusion criteria are met, 3.) the rescheduled date is no more than 14 days past the initial screening date, 4.) the study site is still enrolling subjects]
* have a rash or dermatologic condition or tattoos which may interfere with injection site reaction rating
* have received a blood transfusion or immunoglobulins within 90 days of study entry
* have received a live vaccine within 4 weeks or inactivated vaccine within 2 weeks of study entry
* have previously been vaccinated against influenza for the 2007/2008 northern hemisphere influenza season
* have functional or surgical asplenia
* have a known or suspected problem with alcohol or drug abuse
* were administered an investigational drug within six weeks prior to study entry or are concurrently participating in a clinical study that includes the administration of an investigational product
* are a member of the team conducting this study or are in a dependent relationship with the study investigator. Dependent relationships include close relatives (i.e., children, spouse/partner, siblings, parents) as well as employees of the investigator.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3670 (Actual)
Dates: Start 2007-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Near, MD, Study Director — Baxter Healthcare Corporation
Locations (34):
- United States (34):
  - Tucson, Arizona
  - Anaheim, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Clearwater, Florida
  - Jacksonville, Florida
  - Pembroke Pines, Florida
  - South Miami, Florida
  - Chicago, Illinois
  - Lenexa, Kansas
  - Overland Park, Kansas
  - Lexington, Kentucky
  - Metairie, Louisiana
  - Columbia, Maryland
  - Kansas City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Rochester, New York
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Goose Creek, South Carolina
  - Spartanburg, South Carolina
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Plano, Texas
  - San Angelo, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia

REFERENCES:
- [Derived] Ehrlich HJ, Singer J, Berezuk G, Fritsch S, Aichinger G, Hart MK, El-Amin W, Portsmouth D, Kistner O, Barrett PN. A cell culture-derived influenza vaccine provides consistent protection against infection and reduces the duration and severity of disease in infected individuals. Clin Infect Dis. 2012 Apr;54(7):946-54. doi: 10.1093/cid/cir959. Epub 2012 Jan 19. PMID 22267715
- [Derived] Ehrlich HJ, Berezuk G, Fritsch S, Aichinger G, Singer J, Portsmouth D, Hart MK, El-Amin W, Kistner O, Barrett PN. Clinical development of a Vero cell culture-derived seasonal influenza vaccine. Vaccine. 2012 Jun 19;30(29):4377-86. doi: 10.1016/j.vaccine.2011.11.114. Epub 2011 Dec 13. PMID 22172502
- [Derived] Barrett PN, Berezuk G, Fritsch S, Aichinger G, Hart MK, El-Amin W, Kistner O, Ehrlich HJ. Efficacy, safety, and immunogenicity of a Vero-cell-culture-derived trivalent influenza vaccine: a multicentre, double-blind, randomised, placebo-controlled trial. Lancet. 2011 Feb 26;377(9767):751-9. doi: 10.1016/S0140-6736(10)62228-3. Epub 2011 Feb 15. PMID 21329971

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Influenza Vaccine | Placebo
Started | 1829 | 1841
Completed | 1656 | 1694
Not Completed | 173 | 147

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Influenza Vaccine | Placebo | Total
Number analyzed (Participants) | 1829 | 1841 | 3670
Age, Customized [Count of Participants; unit: Participants]
  ages 18-49 | 1829 | 1841 | 3670
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1037 | 1000 | 2037
  Male | 792 | 841 | 1633
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 315 | 307 | 622
  Not Hispanic or Latino | 1514 | 1534 | 3048
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 15 | 21
  Asian | 33 | 33 | 66
  Native Hawaiian or Other Pacific Islander | 15 | 14 | 29
  Black or African American | 386 | 376 | 762
  White | 1373 | 1388 | 2761
  More than one race | 16 | 15 | 31
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1829 | 1841 | 3670
Weight [Mean (Standard Deviation); unit: kg] | 81.60 (21.104) | 81.87 (20.694) | 81.74 (20.897)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Developing Influenza Infection, as Confirmed by Viral Culture and Typing of Naso-pharyngeal Specimens
Time Frame: 21 days to 180 days after the date of vaccination
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Vaccine | Placebo
Number analyzed (Participants) | 1792 | 1817
Participants | 35 | 62

2. Primary Outcome: The Consistency of Immune Response Produced by 3 Different Lots of VCIV Based on HIA Titer Values
Description: Consistency of each strain across the 3 different lots shown by comparison of the ratios of geometric mean HIA titers at Day 21 between individual lots for the immunogenicity analysis set.
Time Frame: 21 Days after vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titers
Groups:
- Influenza Vaccine Lot 2 vs Lot 1; Influenza Vaccine Lot 3 vs Lot 1; Influenza Vaccine Lot 3 vs Lot 2: Vero-cell derived influenza vaccine
  Inactivated seasonal influenza vaccine (split virus, Vero cell-derived): Trivalent, non-adjuvanted vaccine; dose: 0.5 ml
Arm/Group | Influenza Vaccine Lot 2 vs Lot 1 | Influenza Vaccine Lot 3 vs Lot 1 | Influenza Vaccine Lot 3 vs Lot 2
Number analyzed (Participants) | 569 | 573 | 566
Geometric Mean Titers
  Strain A/H1N1 | 1.22 [1.07 to 1.39] | 1.10 [0.96 to 1.25] | 0.90 [0.79 to 1.02]
  Strain A/H3N2 | 0.94 [0.83 to 1.07] | 0.99 [0.87 to 1.13] | 1.05 [0.93 to 1.20]
  Strain B | 0.88 [0.78 to 0.99] | 0.91 [0.81 to 1.02] | 1.04 [0.92 to 1.17]

3. Secondary Outcome: Frequency and Severity of Occurrence of Any Injection Site Reactions and Systemic Reactions/Adverse Events Related to Vaccination
Time Frame: During the entire 180-day follow-up period
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Vaccine | Placebo
Number analyzed (Participants) | 1829 | 1841
Participants
  Non-Serious Local Reactions: No Reactions | 868 | 1586
  Non-Serious Local Reactions: Mild | 834 | 237
  Non-Serious Local Reactions: Moderate | 99 | 7
  Non-Serious Local Reactions: Severe | 5 | 0
  Non-Serious Local Reactions: Unknown | 23 | 11
  Non-Serious Systemic Reactions: No Reactions | 1199 | 1442
  Non-Serious Systemic Reactions: Mild | 406 | 251
  Non-Serious Systemic Reactions: Moderate | 190 | 132
  Non-Serious Systemic Reactions: Severe | 34 | 16
  Non-Serious Systemic Reactions: Unknown | 0 | 0

ADVERSE EVENTS:
Time Frame: adverse events were recorded during the entire 180-day follow-up period
Arm/Group | Influenza Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 1/1829 | 0/1841
Serious Adverse Events (participants affected / at risk) | 3/1829 | 0/1841
Other Adverse Events (participants affected / at risk) | 1132/1829 | 375/1841
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Influenza Vaccine (N=1829) | Placebo (N=1841)
Death (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — one subject died as a result of a massive open head trauma due to a single motorcycle collision
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) — allergic reaction during administration of investigational product
Acute disseminated encephalomyelitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — subject developed injection site reaction, tingling, burning, itching and numbness after administration of investigational product
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Influenza Vaccine (N=1829) | Placebo (N=1841)
tenderness (Skin and subcutaneous tissue disorders) | 848 | 200
injection site pain (Skin and subcutaneous tissue disorders) | 598 | 140
headache (General disorders) | 327 | 0
muscle pain (Skin and subcutaneous tissue disorders) | 275 | 99
fatigue (General disorders) | 194 | 116
malaise (General disorders) | 137 | 0
shivering (General disorders) | 101 | 0
joint pain (Musculoskeletal and connective tissue disorders) | 96 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less